CLINICAL TRIAL: NCT04959916
Title: Group-Based Metacognitive Therapy for Anxiety and Mood Symptoms in Burns and Plastics Patients: A Feasibility and Acceptability Study
Brief Title: Group-based Metacognitive Therapy for Burns and Plastics Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manchester (Other)
Collaborators: Greater Manchester Mental Health NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Adrian Wells, Professor Adrian Wells, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRAS ID: 287367
Record Dates: First submitted 2021-06-15; First posted 2021-07-13 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Anxiety; Low Mood
MeSH Terms: conditions — Anxiety Disorders; Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: This is a benchmark study, whereby a single group will receive the Group-MCT intervention and this group will be compared to (i.e benchmarked against) data from patients who completed 'Treatment as Usual' within the service.
  The treatment as usual data is collected in the course of normal care. Patients personally identifiable information will be removed from the data base before being shared with the study team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Meta-Cognitive Therapy (Experimental): Group Meta-Cognitive Therapy (Group-MCT)
  Interventions: Behavioral: Group Metacognitive Therapy

INTERVENTIONS:
Behavioral: Group Metacognitive Therapy — Group Meta-Cognitive Therapy (Group-MCT) will consist of six weekly sessions delivered by two trained trainee clinical psychologists over 1-1.5 hours. The aims of the intervention are to help participants develop knowledge that can facilitate control of worry, rumination and attention, and to modify the metacognitive beliefs that maintain these unhelpful patterns of thinking. The treatment follows a manual that has been previously evaluated in the treatment of cardiac patients suffering from anxiety and depression. Sessions include group discussions, experiential learning and homework tasks that participants will be expected to complete between sessions.

SUMMARY:
Serious burns and other traumatic or disfiguring injuries represent a significant public health burden. Survivors often need intense medical or surgical treatment, including plastic surgery. As well as devastating physical injuries, up to 45% of people develop significant mental health difficulties following a traumatic injury. These difficulties include depression, anxiety and post-traumatic stress disorder (PTSD).

Cognitive Behavioural Therapy (CBT) is the most widely offered treatment within the National Health Service (NHS) and the most common treatment provided for burns and plastics patients. However, CBT is limited in efficacy, time-consuming, and focuses on treating the most distressing problem first.

One way to overcome these limitations is to evaluate a group therapy that can treat multiple mental health problems at once. One such treatment is called Metacognitive Therapy (MCT; Wells 2009). MCT targets metacognitive beliefs (beliefs people hold about their thinking) rather than the content of patients' thoughts (i.e. reality testing), which is advantageous over cognitive therapies as often following a burns or plastics injury patients experience realistic negative thoughts (e.g. thoughts about disfigurement). MCT has been shown to be more effective at treating anxiety and depression in mental health settings than CBT, however, more research is needed to evaluate MCT in physical health settings.

The aim of this study is to examine the acceptability and feasibility of group-MCT within the Department of Burns, Plastics and Reconstructive Surgery at Wythenshawe Hospital. We aim to recruit 20 patients to receive six weekly sessions of group-MCT. Sessions will last approximately 90 minutes. Indicators of feasibility and acceptability will be described including rates of referrals, recruitment, and dropout. Data on symptom outcomes (as measured by the PHQ-9 and GAD-7) at pre and post treatment will be assessed and benchmarked against usual treatment delivered. The data will be used to inform a future large-scale trial on the effectiveness of MCT.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients at the Adult Burns Centre in Wythenshawe Hospital;
* Age 18 or older;
* At least one month since the occurrence of the injury;
* A competent level of English language skills (able to read, understand and complete questionnaires in English).
* In the event that sessions will be conducted remotely, participants will require adequate internet connection and access to Microsoft Teams/Zoom.

Exclusion Criteria:

* Cognitive impairment which precludes informed consent or ability to participate;
* Acute suicidality;
* Active psychotic disorders;
* Current drug or alcohol abuse;
* Individuals engaging in active deliberate self-harm;
* Dementia or learning difficulties;
* Antidepressant or anxiolytic medications initiated in the previous 8 weeks;
* Individuals who intentionally set themselves on fire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility indicators | Up to 7 months follow up
  Indicators of feasibility of the group-MCT intervention will be described. Specifically, we will describe rates of:
  * Referrals - the average number of potential patients that are referred to the study per month
  * Recruitment -the average number of patients that meet inclusion, exclusion criteria and that consent to take part in the study, per month.
  * Attendance - Participants will be classified as 'attended', if they attend a minimum of four out of the six group-MCT sessions.
  * Retention - Participants will be classified as 'retained' if they complete the primary symptom measures (GAD-7 and PHQ-9) at the final follow up. Minimal target criteria for retention is 80% of those recruited completing the study.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9; Spitzer et al., 1999). | Administered at baseline, 4 month follow up and 7 month follow up,
  The Patient Health Questionnaire (PHQ-9) is a 9-item questionnaire that wherein individuals rate the frequency at which they experience symptoms of depression from "0" (not at all) to "3" (nearly every day). Total scores can range from 0 - 21, with higher scores indicating higher depression symptoms (i.e., worse outcome)
  *The measure is routinely administered within the service and will be used to benchmark group-MCT against.
Change in Generalized Anxiety Disorder 7-item (GAD-7; Spitzer et al., 2006) scale | Administered at baseline, 4 month follow up and 7 month follow up,
  The Generalized Anxiety Disorder 7-item (GAD-7) is a 7-item screening tool that measures common symptoms of anxiety. Total scores can range from 0 - 21, with higher scores indicating higher anxiety (i.e., worse outcome)
  *The measure is routinely administered within the service and will be used to benchmark group-MCT against.
Change in Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983) | Administered at baseline, 4 month follow up and 7 month follow up,
  The Hospital Anxiety and Depression Scale (HADS) is a brief 14-item self-report measure of anxiety and depression symptoms. Total scores for depression and anxiety can range from 0 - 21, with higher scores indicating higher symptoms of anxiety/depression (i.e., worse outcome).
Change in Metacognitions Questionnaire (MCQ-30; Wells & Cartwright-Hatton, 2004). | Administered at baseline, 4 month follow up and 7 month follow up,
  The Metacognitions Questionnaire (MCQ-30) is a 30-item self-report measure assessing metacognitive beliefs. Total score can range from 0 - 120, with a higher score indicating worse outcome.
Change in Impact of Event Scale-Revised (IES-R; Weiss & Marmar, 1997). | Administered at baseline, 4 month follow up and 7 month follow up,
  The Impact of Event Scale-Revised (IES-R) is a 22-item self-report measure that assesses subjective distress caused by traumatic events. Total score ranges from 0 - 88 and higher scores indicate worse trauma symptoms (i.e., worse outcome).
Change in Beliefs About Memory Questionnaire (BAMQ; Bennett & Wells, 2010). | Administered at baseline, 4 month follow up and 7 month follow up,
  The Beliefs About Memory Questionnaire (BAMQ) is a 15-item scale that measures positive and negative beliefs about trauma memory. Scores can range from 0 - 60, higher scores are considered worse outcomes.
Change in Cognitive Attentional Syndrome Scale 1 Revised (CAS-1R; Wells, 2015) | This will be administered to track any changes in participants' metacognitive beliefs, knowledge or strategies. It will be administered at every group-MCT intervention session (i.e. group-MCT sessions 1, 2, 3, 4, 5 and 6).
  This measure assesses a perseverative thinking style that contributes to and maintains emotional distress in the meta-cognitive model (e.g., worry/rumination and other coping strategies, and metacognitive beliefs). Scores can range from 0-1000 and higher scores are considered worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Burns Plastics and Reconstructive Surgery, Wythenshawe Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data may be used for future research at the discretion of the data custodian as long as the data being used is not identifiable and is not combined with any other data which makes it identifiable. Data will only be shared in line with what has been agreed in the informed consent process.

REFERENCES:
- [Background] Wells, A. (2009). Metacognitive therapy for anxiety and depression. New York: Guilford press.
- [Background] Davydow DS, Katon WJ, Zatzick DF. Psychiatric morbidity and functional impairments in survivors of burns, traumatic injuries, and ICU stays for other critical illnesses: a review of the literature. Int Rev Psychiatry. 2009 Dec;21(6):531-8. doi: 10.3109/09540260903343877. PMID 19919206